CLINICAL TRIAL: NCT04650958
Title: Subthalamic Nucleus Deep Brain Stimulation in Isolated Generalized or Segmental Dystonia: A Multicenter, Randomized, Double-blind, Sham-controlled, Parallel-group Trial
Brief Title: SUNDYS: A Multicenter, Randomized, Double-blind, Sham-controlled, Parallel-group Trial
Acronym: SUNDYS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Collaborators: Renmin Hospital of Wuhan University (Other); Shanghai Tongji Hospital, Tongji University School of Medicine (Other); Second Affiliated Hospital of Soochow University (Other); West China Hospital (Other)
Responsible Party: Principal Investigator, Bomin Sun, Director of Center for Functional Neurosurgery, Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Ruijin_SUNDYS
Record Dates: First submitted 2020-11-19; First posted 2020-12-03 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Dystonia
Keywords: Deep brain stimulation; Subthalamic nucleus; Randomized controlled trial
MeSH Terms: conditions — Dystonia | interventions — Deep Brain Stimulation

STUDY DESIGN:
Intervention Model Description: In this study after having DBS leads implanted successfully, 38 patients will be randomly assigned to either the control or experimental group with a 1:1 allocation. The experimental group will receive continuous DBS stimulation for 3 months, while controls will have sham stimulation for 3 months.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The randomization will be conducted by the Coordination Center of Clinical Trials (CenTrial) in order to keep the researchers managing the data and the statistician blind to group assignment and the study conditions. All the clinical assessments done during the trial period will be double-blind, e.g., neither the patient not the clinician or study personnel involved in the scoring will not be aware of the condition of stimulation. All personnel, except the physician-programmer responsible for the DBS setting, will be blinded to the identity of the parameters. While programming the programmer will not sit face-to-face with the patient, but in another room adjusting the parameter wirelessly with the help of the attending doctor who will inform the programmer of the patient's reaction. The electrical parameters will be tested in all patients which means they all will perceive similar stimulation related sensations during each follow-up.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STN DBS stimulation group (Active Comparator): In the STN DBS stimulation group, patients will receive a continuous DBS stimulation for 3 months and the first default parameters applied will be monopolar setting (0.5 V under threshold that causes side effects, 135 Hz, 90 µs, at one of the two dorsal contacts). If the default parameters are found not suitable for an individual patient due to unexpected reasons, an alternative method will be applied (e.g., decreased voltage) to try to maintain full compliance with the scheduled study.
  Interventions: Procedure: Deep brain stimulation
- Sham stimulation group (Sham Comparator): In the sham stimulation group, the programming will also start within 1 week after the surgery, but at each follow-up the DBS system will be turned off after the parameter is adjusted to the threshold that causes side effects without continuous stimulation. After the 3-month double-blind period the patients can choose to set on the DBS system again and receive regular continuous stimulation treatment.
  Interventions: Procedure: Deep brain stimulation

INTERVENTIONS:
Procedure: Deep brain stimulation — Deep brain stimulation (DBS) has been in use to treat patients with movement disorders since 1989, with many thousands of publications showing its effectiveness. DBS for dystonia received the US FDA mark in 2003 and China FDA mark in 2016. In this study, the DBS system devices are manufactured and donated by SceneRay (Suzhou, China). The Stimulator System is implanted by a qualified neurosurgeon and consists of three implantable components: the leads, the extension wires and the neurostimulator. The DBS programming will start within 1 week after the surgery completed.

SUMMARY:
Dystonia is a group of movement disorders characterized by twisting, repetitive movements, or abnormal postures caused by involuntary muscle contractions and is characterized by a young age of onset and a high disability rate. Early intervention can reduce disability incidence, improve the patient's quality of life, and reduce the burden on families and society. Multiple international guidelines on dystonia have found deep brain stimulation (DBS) to be a safe and effective treatment for refractory dystonia. The globus pallidal internus (GPi) is the mostly widely used target for dystonia. However, there are limitations on the GPi DBS treatment, including slow onset of beneficial effects, poor improvement of axis symptoms, and potential stimulation-related side effects. Previous studies have described the highly successful use of subthalamic nucleus deep brain stimulation (STN DBS) in patients with refractory dystonia, suggesting that STN DBS is an effective and persisting alternative to pallidal deep brain stimulation. However, all STN DBS treated cases have been analyzed in open-label uncontrolled cohort studies, leading to limited data with a high level of evidence on the STN DBS in dystonia. Further, the investigators hypothesized STN has potentially more effectiveness when compared with GPi, and may be more power-saving and quick-acting. In this study, the investigators will organize a prospective randomized, double-blind, parallel-group, multicenter study comparing active versus sham stimulation in isolated segmental or generalized dystonia to evaluate the effectiveness and safety of STN DBS by measuring the impact on motor status, mental status, quality of life, the rate of response of the patients (the number of patients with ≥30% improvement in the movement score on the Burke-Fahn-Marsden Dystonia Rating Scale) and the rate of adverse events during the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must meet criteria for the diagnosis of isolated generalized or segmental dystonia, including idiopathic and inherited dystonia, as defined by the Phenomenology and Classification of Dystonia: A Consensus Update 2013;
2. Patients will be ≥ 14 years old;
3. The course of disease will be ≥ 3 years;
4. Patients will have:

   1. Significant dystonia symptoms;
   2. Compromised life quality;
   3. Unsatisfactory response to oral treatment with anticholinergic agents antiepileptic agents, anti-dopamine agents, dopaminergic agents, or muscle relaxants;
   4. Unsatisfactory response to or contraindication for previous botulinum toxin treatment; and
   5. Ability to provide written informed consent.

Exclusion Criteria:

1. Patients with a diagnosis or probable diagnosis of acquired, compound, and complex dystonia, as defined by the Phenomenology and Classification of Dystonia: A Consensus Update 2013;
2. Previous brain surgery for dystonia;
3. Patients with cognitive impairment (MMSE score <24) or moderate-severe depressive disorder (BDI>25);
4. Patients with marked brain atrophy identified by magnetic resonance imaging (MRI) or computed tomography (CT);
5. Patients with other medical or psychiatric comorbidities that could increase the surgical risk or interfere with completion of the trial;
6. Patients with increased bleeding risk, or other factors contraindicating neurosurgery or general anesthesia;
7. Patients unable to cooperate with the assessments during the follow-up.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
The change from baseline to 3 months after stimulation of Burke-Fahn-Marsden Dystonia Rating Scale (BFMDRS) score | Baseline; 3months after stimulation
  The scale consists of a movement and disability subscale with scores ranging from 0 to 120 and 0 to 30, respectively, higher scores indicating greater impairment.

SECONDARY OUTCOMES:
Abnormal Involuntary Movement Scale (AIMS) | Baseline; 1 week, 1 month and 3months after stimulation
  The AIMS is a 12-item clinician-rated scale to assess severity of dyskinesias. These items are rated on a five-point scale of severity from 0-4. The scale is rated from 0 (none), 1 (minimal), 2 (mild), 3 (moderate), 4 (severe). Two of the 12 items refer to dental care.
36-item Short-Form General Health survey (SF-36) | Baseline; 1 week, 1 month and 3months after stimulation
  SF-36 is a measure of health-related quality-of-life with a 36-item patient-reported questionnaire that covers eight health domains. Higher scores indicate a more favorable health state.
Beck Depression Inventory-II (BDI) | Baseline; 1 week, 1 month and 3months after stimulation
  BDI contains 21 questions, each answer being scored on a scale value of 0 to 3. Higher total scores indicate more severe depressive symptoms.
Beck Anxiety Inventory (BAI) | Baseline; 1 week, 1 month and 3months after stimulation
  BAI contains 21 questions, each answer being scored on a scale value of 0 to 3. Higher total scores indicate more severe anxiety symptoms.
Montreal Cognitive Assessment (MoCA) | Baseline; 3months after stimulation
  MoCA scores range between 0 and 30. A score of 26 or over is considered to be normal. Lower scores indicate more disability.
Cambridge Neuropsychological Test Automated Battery (CANTAB) | Baseline; 3months after stimulation
  A detailed computerized cognitive battery selected from CANTAB includes: Stockings of Cambridge (SOC) and Spatial working memory (SWM) for executive function; Motor screening task (MOT) and a five-choice series selection task for attention; Paired associates learning (PAL) and Pattern recognition memory (PRM) for memory.
The rate of response | 1 week, 1 month and 3months after stimulation
  The number of patients with ≥30% improvement in the movement score on the BFMDRS
The rate of adverse event (AE) | Within 1 week after surgery; 1 week, 1 month and 3months after stimulation
Burke-Fahn-Marsden Dystonia Rating Scale (BFMDRS) | 1 week and 1 month after stimulation
  The scale consists of a movement and disability subscale with scores ranging from 0 to 120 and 0 to 30, respectively, higher scores indicating greater impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Bomin Sun, Principal Investigator — Ruijin Hospital
Locations (1):
- Shanghai Ruijin Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Hu K, Wu Y, Shen T, Zhou J, Li H, Dong H, Yi W, Luo C, Jin L, Liu C, Shang H, Zhan S, Li D, Wu Y, Benabid AL, Sun B; SUNDYS investigators. Effectiveness and safety of subthalamic nucleus deep brain stimulation in isolated generalised or segmental dystonia (SUNDYS trial): a study protocol. Br J Neurosurg. 2025 Sep 22:1-9. doi: 10.1080/02688697.2025.2562277. Online ahead of print. PMID 40981502